CLINICAL TRIAL: NCT02424370
Title: Geriatric Evaluation to Predict Mortality and Functional Recovery After Trans Aortic Valve Implantation. Multicenter Observational Study
Brief Title: Geriatric Evaluation to Predict Mortality and Functional Recovery After Trans Aortic Valve Implantation
Acronym: EVA-G-TAVI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: NI11069
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-03

CONDITIONS: Symptomatic Aortic Stenosis
Keywords: Aortic stenosis; TAVR; Frailty; Elderly
MeSH Terms: conditions — Aortic Valve Stenosis; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: TAVR — Percutaneous aortic valve replacement
  Other Names: Trans-aortic Valve Replacement

SUMMARY:
Transcutaneous trans-aortic valve replacement (TAVR) is now a common procedure to treat symptomatic aortic stenosis. Although as effective and safe as surgical aortic valve replacement, it is still restricted to high surgical risk patient who are frail. The aim of the TAVI-EVA is to identify geriatric biomarkers that may help to predict survival and functional recovery after TAVR

DETAILED DESCRIPTION:
Primary objective: identify geriatric biomarkers associated with vital/functional status after TAVR.

Primary outcome measure is altered functional status at six month follow-up defined as an absolute decrease of 15 points of the Barthel Index.

Secondary outcome measures are: Barthel index and survival at 6, 9 and 12 months follow-up. QOL during follow-up

ELIGIBILITY:
Inclusion Criteria:

* Age ≥75
* Symptomatic aortic stenosis
* Prior geriatric evaluation
* Patient who agreed to answer the telephone follow-up to 6, 9 and 12 months
* Patient given his non-opposition to using his data
* Patient affiliated to the French social security.

Exclusion criteria:

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: person aged over 75 years with indication for implantation of TAVI
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Maintaining or improving the level of functional independence, defined as a score of Barthel index at 6 months | at 6 months

SECONDARY OUTCOMES:
Score of Barthel | at 6, 9 and 12 months
  Maintaining of the same Score
Maintain or improve the quality of life score at 6 months, defined as a score of SF-12 scale at 6 months | at 6 months
Survival rate at 6 months, 9 months, 12 months | at 6, 9 and 12 months
Survival time after TAVI during the study | up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Joël BELMIN, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Jean Philippe COLLET, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Institut de Cardiologie-GH Pitié Salpétirère, Paris, Île-de-France Region, France